CLINICAL TRIAL: NCT01526824
Title: The Effects of Polyunsaturated Omega-3 Fatty Acids (Lovaza) on Patients Taking Clopidogrel +/- Aspirin Who Have Suffered an Ischemic Stroke/TIA and/or Are Candidates for Neuroendovascular Stenting.
Brief Title: Lovaza's Effect on Clopidogrel in a Neuro Population
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Millard Fillmore Gates Hospital (Other)
Collaborators: Kaleida Health (Other)
Responsible Party: Principal Investigator, Melissa Baxter, Neuroscience Clinical Pharmacy Coordinator, Millard Fillmore Gates Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHP1061010A
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Docosahexaenoic Acids; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm, clopidogrel without Lovaza (No Intervention): These patients will be receiving standard of care therapy with either standard dose (75mg daily) or high dose (150mg daily) clopidogrel +/- aspirin based on physician discretion.
- Clopidogrel plus Lovaza (Experimental): This is the study arm of the trial, in which patients will be receiving either a standard dose (75mg daily) or high dose (150mg daily) clopidogrel with or without aspirin as well as therapy with daily Lovaza.
  Interventions: Dietary Supplement: omega-3 polyunsaturated fatty acids (Lovaza)

INTERVENTIONS:
Dietary Supplement: omega-3 polyunsaturated fatty acids (Lovaza) — Lovaza, 1 gram orally daily
  Arms: Clopidogrel plus Lovaza

SUMMARY:
In patients who have suffered an ischemic stroke or TIA (mini-stroke), as well as in patients who are candidates for neuroendovascular stenting, it is standard of care to treat these patients with antiplatelet therapy, or "blood-thinners", the most common of which is clopidogrel (Plavix) with or without the addition of aspirin. A relatively common problem encountered with these patients is non-responsiveness to clopidogrel therapy. A prior study in cardiac patients showed that the addition of omega-3 polyunsaturated fatty acids (Lovaza, or "fish oil") can increase a patient's response to therapy with clopidogrel, but there have been no studies in neuro patients. In this study, patients will be divided into one of two groups: in the study arm, patients will receive clopidogrel +/- aspirin as well as Lovaza. In the control arm, patients will only receive clopidogrel +/- aspirin. Assays will be done to measure responsiveness to clopdiogrel on days 0, 12-24 hours after loading dose, day 3-5 if still inpatient, and at a follow-up visit 20-30 days after the start of the study. The investigators believe that this study will show an increase in platelet aggregation in patients receiving both clopidogrel and Lovaza.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male and female
* Age range: 25 - 80 years of age
* Study population: Patients who require antiplatelet therapy with clopidogrel +/- aspirin who are candidates for neuroendovascular stenting or have had an ischemic stroke/TIA.
* Eligible females will be: Non-pregnant nor lactating/breastfeeding; Be surgically sterile for at least 6 months, postmenopausal, or if heterosexually active and of childbearing potential, agree to continue to use an accepted method of birth control throughout the study.

Exclusion Criteria:

* Any clinically significant abnormal finding uncovered during the physical examination and/or clinically significant abnormal laboratory result at screening according to the clinical judgment of the Investigators
* Current alcohol abuse
* Smokers unable to refrain from smoking during the clinical trial
* Patients who are already taking anticoagulants or other antiplatelets (ticlopidine, prasugrel, dipyridamole, cilostazol), or patients already taking PUFAs
* Patients taking medications known to interact with clopidogrel that cannot be held or changed due to increased risk of adverse health events.

  * Cytochrome P450 3A4 and 2C19 (CYP3A4, CYP2C19) inhibitors or substrates known to cause competitive inhibition
  * Proton pump inhibitors (PPIs)
  * NSAIDs
* Pregnant women or lactating/breastfeeding women.
* Active or recent major bleeding (within 14 days) using TIMI score (minor severity will be acceptable based on clinical examination/patient history)

  * Major severity-
* Intracranial hemorrhage
* Cardiac tamponade
* Overt bleeding with a decrease in hemoglobin ≥ 5 g/dl or a decrease in hematocrit ≥ 15% (with or without an identifiable site)

  * Minor severity-
* Spontaneous gross hematuria
* Spontaneous hematemesis
* Spontaneous hemoptysis
* Observed bleeding with decrease in hemoglobin ≥ 3 g/dl but ≤ 5 g/dl (with an identifiable site)
* History of gastric or duodenal ulcer
* Platelet count < 100 x 109/L
* Serum creatinine > 2 mg/dL
* Liver injury (alanine transaminase level > 1.5 times upper limit of normal)
* Recent surgery (within 14 days of study screening)
* Known bleeding diathesis including but not limited to

  * Hemophilia
  * Von Willebrand disease
  * Leukemia
  * Clotting factor deficiencies
* Uncontrolled hypertension

  * Sustained systolic blood pressure > 185 mmHg, despite treatment
  * Sustained diastolic blood pressure > 110 mmHg, despite treatment
* Hypersensitivity or intolerance to clopidogrel, aspirin, PUFAs and/or documented fish allergy
* Patients who are currently enrolled in a different study or who have taken an investigational medication 30 days prior to starting this study.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
PRU and % inhibition of P2Y12 Assay | 20-30 days after initiation of the study

SECONDARY OUTCOMES:
Neurologic events in each study | 20-30 days after initiation of study
HDL, triglycerides, LDL, or total cholesterol | 20-30 days after initiation of the study
Bleeding | 20-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Baxter, PharmD, Principal Investigator — Millmore Fillmore Gates Hospital
Locations (1):
- Millmore Fillmore Gates Hospital, Buffalo, New York, United States